CLINICAL TRIAL: NCT00141349
Title: A Double-Blind, Placebo Controlled, Parallel Group, Multicenter Study to Assess the Time to Onset, Safety, and Toleration of Differing Doses and Combinations of Immediate Release and Modified Release Formulations of UK369,003 in Adult Male Subject With Erectile Dysfunction
Brief Title: Assessment of Onset, Safety & Toleration of UK-369,003 in Male Erectile Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3711029
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2006-07-25 (Estimated); Status verified 2006-01

CONDITIONS: Impotence
MeSH Terms: conditions — Erectile Dysfunction | interventions — 1-(6-ethoxy-5-(3-ethyl-6,7-dihydro-2-(2-methoxyethyl)-7-oxo-2H-pyrazolo(4,3-d)pyrimidin-5-yl)-3-pyridyl sulphonyl)-4-ethylpiperazine

INTERVENTIONS:
Drug: UK-369,003

SUMMARY:
To determine the onset of action, safety and toleration of different formulations and doses of UK-369,003 in patients with erectile dysfunction. Patients should have been previously treated with PDE5 inhibitors and have been responders to the drugs. Duration of treatment is 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Erectile dysfunction as defined by DSM-IV. Patients should have been PDE5 inhibitor respondents

Exclusion Criteria:

* Alpha blockers and Nitrates of any preparation

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-02; Study Completion 2005-08

PRIMARY OUTCOMES:
The time needed to obtain an erection hard enough to attempt sexual intercourse.

SECONDARY OUTCOMES:
Proportion of responders based on successful erections Based on erections hard enough for sexual intercourse 15, 45 and 60 minutes post dose Proportion of good responders based on successful erections International Index of Erectile Function

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (33):
- United States (33):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Tempe, Arizona
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, San Bernardino, California
  - Pfizer Investigational Site, Torrance, California
  - Pfizer Investigational Site, Waterbury, Connecticut
  - Pfizer Investigational Site, Aventura, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Fort Wayne, Indiana
  - Pfizer Investigational Site, Jeffersonville, Indiana
  - Pfizer Investigational Site, Metairie, Louisiana
  - Pfizer Investigational Site, Milford, Massachusetts
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Endwell, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Beachwood, Ohio
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Bryan, Texas
  - Pfizer Investigational Site, Sugar Land, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, West Jordan, Utah
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Milwaukee, Wisconsin